CLINICAL TRIAL: NCT01211691
Title: Study of the Anti-EphA3 Monoclonal Antibody KB004 in Subjects With EphA3-Expressing Hematologic Malignancies
Brief Title: Study of KB004 in Subjects With Hematologic Malignancies (Myelodysplastic Syndrome, MDS, Myelofibrosis, MF)
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: KaloBios to Wind Down Operations
Sponsor: Humanigen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB004-01
Record Dates: First submitted 2010-09-24; First posted 2010-09-29 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Myelodysplastic Syndrome (MDS); Myelofibrosis (MF)
Keywords: Hematologic; Leukemia; Malignancies; Myeloproliferative Neoplasms
MeSH Terms: conditions — Myelodysplastic Syndromes; Primary Myelofibrosis; Leukemia; Neoplasms; Myeloproliferative Disorders | interventions — KB004

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase 1 dose levels: KB004 (Experimental): IV infusion 1x Weekly for a 21 day dosing cycle
  Subjects with heme malignancies will be assigned to one of 11 planned KB004 (dose levels (20mg, 40mg, 70mg, 100mg, 140mg, 190mg, 250mg, 330mg)
  Interventions: Drug: KB004, Monoclonal Antibody
- Phase 2 dose levels: KB004 (Experimental): IV infusion 1x Weekly for a 21 day dosing cycle
  Subjects will be assigned to the recommended Phase 2 dose of 250 mg
  Interventions: Drug: KB004, Monoclonal Antibody

INTERVENTIONS:
Drug: KB004, Monoclonal Antibody

SUMMARY:
This is a global, multicenter, open-label, repeat-dose, Phase 1/2 study consisting of a Dose Escalation Phase (Phase 1) and a Cohort Expansion Phase (Phase 2). In both phases, KB004 will be administered by IV infusion once weekly as part of a 21-day dosing cycle.

DETAILED DESCRIPTION:
The purpose of Phase 1 is to determine a maximum tolerated dose (MTD) for KB004 when administered to subjects with hematologic malignancies who meet the entry criteria. Phase 1 has completed enrollment July of 2014, the recommended Phase 2 dose is 250 mg. AML 20 mg Cohort completed enrollment Dec 2014.

The purpose of Phase 2 is to characterize preliminary clinical activity. The Phase 2 portion of the study consists of two parts:

* Part A: Subjects with AML or MDS who meet the entry criteria
* Part B: Subjects with MF who meet the entry criteria

ELIGIBILITY:
Key Inclusion Criteria (Phase 1):

- Confirmed hematologic malignancy, including Acute Myeloid Leukemia (AML), Chronic Lymphocytic Leukemia (CLL), Chronic Myelogenous Leukemia (CML), Acute Lymphocytic Leukemia (ALL), Myelodysplastic Syndrome (MDS), Multiple Myeloma (MM), Myelofibrosis (MF), Myeloproliferative Neoplasms (MPN) or MDS/MPN overlap diseases. (Once Phase 2 has started subjects with AML will be eligible for inclusion in the Phase 1 portion of the study only if their malignancy has been shown to have c-Cbl mutation, trisomy 3, trisomy 11, inv(16), or elevated FLT3. [Other AML and subjects with MDS will no longer be eligible for inclusion in the Phase 1 portion of the study]).

Key Inclusion Criteria (Phase 2):

* Part A: AML or MDS patients with an acceptable level of EphA3 expression
* Part B: MF patients with an acceptable level of EphA3 expression

Key Inclusion Criteria (Both Phases):

* Confirmed hematologic malignancy refractory to or progressed following standard treatments, or subjects not considered medically suitable to receive standard of care treatment or who refuse standard of care treatment
* Acceptable level of EphA3 expression
* Eastern Cooperative Oncology Group (ECOG) ≤1
* Acceptable laboratory results

Key Exclusion Criteria (Both Phases):

* For subjects with AML, more than 2 prior therapies for AML (induction and consolidation with or without a hypomethylating agent given in a maintenance setting are considered 1 therapy)
* History of or current central nervous system (CNS) involvement that may increase risk of bleeding
* Recent major surgery
* Ongoing surgical or wound healing complications
* Active clinically significant bleeding
* Uncontrolled hypertension
* Significant intercurrent illness
* Known history of prolonged bleeding times or platelet dysfunction
* Active infection requiring IV antibiotics, IV antifungals, or IV antivirals within 2 weeks prior to Cycle 1, Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-09; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Determine a possible maximum tolerated dose (MTD) | Once weekly for the first three weeks of study treatment
Phase 2: To characterize preliminary clinical activity based on the International Working Group (IWG) criteria specific to the hematologic malignancy | Evaluations at designated timepoints

SECONDARY OUTCOMES:
Phase 1: Examine clinical activity | Evaluations at designated timepoints
Phase 1/2: Safety and Tolerability | Duration of study participation
Phase 1/2: Pharmacokinetic profile | Cycle 1: multiple timepoints. Thereafter, single samples at designated cycles
Phase 1/2: Assess immunogenicity | Cycle 1: multiple timepoints. Thereafter, single samples at designated cycles

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Lam, Study Director — Humanigen, Inc.
Locations (9):
- United States (7):
  - Palo Alto, California
  - Sacramento, California
  - Miami, Florida
  - Tampa, Florida
  - Manhattan, New York
  - Cleveland, Ohio
  - Houston, Texas
- Australia (2):
  - Adelaide, South Australia
  - Prahran, Victoria

REFERENCES:
- [Derived] Swords RT, Greenberg PL, Wei AH, Durrant S, Advani AS, Hertzberg MS, Jonas BA, Lewis ID, Rivera G, Gratzinger D, Fan AC, Felsher DW, Cortes JE, Watts JM, Yarranton GT, Walling JM, Lancet JE. KB004, a first in class monoclonal antibody targeting the receptor tyrosine kinase EphA3, in patients with advanced hematologic malignancies: Results from a phase 1 study. Leuk Res. 2016 Nov;50:123-131. doi: 10.1016/j.leukres.2016.09.012. Epub 2016 Sep 28. PMID 27736729